CLINICAL TRIAL: NCT06397235
Title: DEB-TACE in Combination With or Without RALOX-based HAIC for Unresectable Large Hepatocellular Carcinoma: A Randomized, Controlled Trial
Brief Title: DEB-TACE+RALOX-HAIC vs DEB-TACE for Large HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other); Guangzhou Development District Hospital (Unknown); The Affiliated Shunde Hospital of Jinan University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-19
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; transarterial chemoembolization; drug-eluting beads; hepatic artery infusion chemotherapy; oxaliplatin; raltitrexe
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB-TACE+HAIC (Experimental): For DEB-TACE, superselective catheterization is performed and CalliSpheres loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In patients with huge or bilobar multiple lesions, in order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session.
  After each chemoembolization, the microcatheter is reserved at the main hepatic tumor-feeding artery. The RALOX-based regimen is intra-arterially administered.
  During follow-up, the treatment will be repeated on demand (about 4-week interval) based on the evaluation of the follow-up laboratory and imaging examination.
  Interventions: Drug: DEB-TACE+HAIC
- DEB-TACE (Active Comparator): Superselective catheterization is performed and CalliSpheres loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In patients with huge or bilobar multiple lesions, in order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session.
  Interventions: Drug: DEB-TACE

INTERVENTIONS:
Drug: DEB-TACE+HAIC — CalliSpheres (100-300 µm) loaded with pirarubicin for transarterial chemombolization: Typically, one vial of the beads was loaded with 60 mg pirarubicin. If blushed tumors is still visible after the embolization with one vial of beads, regular microspheres (8spheres) with diameters of 100-700 μm are additionally injected.
  RALOX-based regimen for hepatic arterial infusion chemotherapy: oxaliplatin, 85 mg/m2 infusion for 2 hours; Raltitrexed, 3 mg/m2 infusion for 0.5 hour.
  Arms: DEB-TACE+HAIC
Drug: DEB-TACE — CalliSpheres (100-300 µm) loaded with pirarubicin for transarterial chemombolization: Typically, one vial of the beads was loaded with 60 mg pirarubicin. If blushed tumors is still visible after the embolization with one vial of beads, regular microspheres (8spheres) with diameters of 100-700 μm are additionally injected.
  Arms: DEB-TACE

SUMMARY:
This study is conducted to evaluate the efficacy and safety of transarterial chemoembolization with drug-eluting beads (DEB-TACE) combined with hepatic artery infusion chemotherapy (HAIC) with oxaliplatin and raltitrexed (RALOX-HAIC) versus DEB-TACE alone for unresectable large hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a multicenter randomized study to evaluate the efficacy and safety of DEB-TACE plus RALOX-HAIC (DEB-TACE+HAIC) compared with DEB-TACE alone for unresectable large HCC (>7cm).

130 patients with unresectable large HCC (> 7cm) will be enrolled in this study. The patients will receive either DEB-TACE+HAIC or DEB-TACE using an 1:1 randomization scheme. In the DEB-TACE+HAIC arm, the microcatheter will be reserved at the main hepatic tumor-feeding artery and chemotherapy drugs (RALOX-based regimen) will be intra-arterially administered though the microcatheter. In the DEB-TACE arm, patients will be treated with DEB-TACE alone. The treatments can be repeated on demand (at a 4-week interval usually) based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team. During follow-up, the potential resectability of the tumor will be assessed by the multidisciplinary team (MDT). Once the tumors become resectable, curative surgical resection will be recommended for the patients.

The primary end point of this study is progression-free survival (PFS). The secondary endpoints are tumor response (objective response rate and disease control rate), overall survival (OS) , and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* HCC confirmed by histology/cytology or diagnosed clinically.
* At least one measurable intrahepatic target lesion.
* The largest tumor size > 7 cm.
* Tumor recurrence after curative treatment (hepatectomy or ablation) is eligible for enrollment.
* Child-Pugh score 5-7.
* ECOG performance status ≤ 1.
* Adequate organ and hematologic function with platelet count ≥75×10^9/L, leukocyte >3.0×10^9/L, Neutrophil count ≥1.5×10^9/L, ASL and AST≤5×ULN, creatinine clearance≤1.5×ULN, and prolongation of prothrombin time ≤4 seconds.

Exclusion Criteria:

* Macrovascular invasion or extrahepatic metastasis.
* Diffuse HCC.
* Decompensated liver function, including: ascites, bleeding from gastroesophageal varices, and hepatic encephalopathy.
* Previous palliative treatments, including TACE, transcatheter arterial embolization, HAIC, radiation therapy, systemic therapy.
* Organ (heart and kidneys) dysfunction, unable to tolerate TACE or HAIC treatment.
* History of other malignancies.
* Uncontrollable infection.
* History of HIV.
* Gastrointestinal bleeding within 30 days, or other bleeding> CTCAE grade 3.
* History of organ or cells transplantation.
* Pregnant or lactating patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST.
Disease control rate (DCR) | 3 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST.
Overall survival (OS) | 4 years
  The time from date of randomization to death due to any cause.
Adverse Events (AEs) | 3 years
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided